CLINICAL TRIAL: NCT03312088
Title: A Prospective, Multi-center, Single Arm Adaptive-design Study to Evaluate the Survivorship of the Maxx Orthopedics' PCK System in Revision Cases
Brief Title: Maxx Orthopedics' PCK Revision TKA Study of Component Survivorship
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maxx Orthopedics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MO-2017-PCK
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Aseptic Loosening; Infection; Bone Loss; MCL - Medial Collateral Ligament Rupture of the Knee; Periprosthetic Fractures
MeSH Terms: conditions — Infections; Bone Diseases, Metabolic; Periprosthetic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Freedom Knee PCK Components — Total Knee Revision

SUMMARY:
The objectives of this clinical investigation are to evaluate the safety and performance of the Freedom Total Knee® PCK System.

DETAILED DESCRIPTION:
The clinical investigation is designed to be prospective to ensure that the population is representative of the type of population for which the Freedom Total Knee® System with the revision components is intended to treat. Subjects with a primary diagnosis of end-stage symptomatic revision knee who require a uni-lateral knee prosthesis and have been evaluated as appropriate candidates for a revision total knee arthroplasty, by the Investigator, will be invited to take part in this clinical investigation. Patients will be drawn from hospital clinics focusing on this type of treatment.

The treatment period of 36 months is considered sufficient to monitor the safety and clinical performance of the device. However, the patients will be contacted annually for 10 years or as long as the patient is willing to monitor their long-term progress.

An interim report will be issued when at least 120 patients will complete the 12-month follow-up.

No treatments will be withheld as part of this clinical investigation although any other treatments that need to be administered during the clinical investigation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 40 years of age or older and less than 80 years of age (>40 and <80 years).
* Patients having undergone a primary TKR and are candidates for a revision surgery based on aseptic loosening, infections, bone loss, MCL disruption, and/or periprosthetic fractures.
* Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and the prescribed rehabilitation.
* Subjects who, in the opinion of the Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.

Exclusion Criteria:

* Primary knee replacement of the affected knee joint
* Other significant disabling problems from the muscular-skeletal system than in the knees (i.e muscular dystrophy, polio, neuropathic joints)
* Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living.
* Patients who are found to be non-compliant by their physician
* Patients with or having; malignancy - active malignancy, active or suspected systemic infection, Paget's disease, renal osteodystrophy, immunologically suppressed, sickle cell anemia, and systemic lupus erythmatosus.
* The patient has a neuromuscular or neurosensory deficit.
* Female patients planning a pregnancy during the course of the study.
* Patients, who are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
* Varus or valgus deformity > 20 degrees
* Bilateral TKR

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having undergone a primary TKR and are candidates for a revision surgery based on aseptic loosening, infections, bone loss, MCL disruption, and/or periprosthetic fractures.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 36 months
  "No Explants"

SECONDARY OUTCOMES:
Revision rates of any component (including insert) for any reason. | 36 months
  Revision rates of any component (including insert) for any reason.
Revision rates of any component (including insert) for any reason except infection. | 36 months
  Revision rates of any component (including insert) for any reason except infection.
KSS | 36 months
  Knee Society Score
WOMAC | 36 months
  Pain Score
ROM | 36 months
  Range of Motion

CONTACTS AND LOCATIONS:
Overall Officials: David Cashin, MD, Principal Investigator — Coastal Orthopedics
Locations (1):
- Coastal Orthopedics, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No